CLINICAL TRIAL: NCT04341805
Title: Application of Hyperoxygenated Fatty Acids in a Surgical Wound of the Umbilical Trocar After Laparoscopic Cholecystectomy With Placement of a Prosthesis in Patients With Risk Factors
Brief Title: Application of Hyperoxygenated Fatty Acids in a Surgical Wound After Laparoscopic Cholecystectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Marta Bellón, Physician, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AGHO-MYL01/2020
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A. Physiological saline. (Active Comparator): The surgical procedure in group A consisted of the placement of a 6.4cm diameter circular prosthesis (BARD Hernia Patch) at the intra-abdominal level. Subsequently, the liquid contained in the 10 ml opaque vial was administered (Ecolav Physiological Washing Serum 0.9%, (SSF).
  Interventions: Procedure: Physiological saline
- Group B. Solution hyperoxygenated fatty acids (Experimental): The surgical procedure in group B consisted of the placement of a 6.4cm diameter circular prosthesis (BARD Hernia Patch) at the intra-abdominal level. Subsequently, the liquid contained in the 10 ml opaque vial (AGHO solution) was administered according to randomization.
  Interventions: Procedure: PrevOmega

INTERVENTIONS:
Procedure: PrevOmega — The intervention consisted of placing a prosthesis at the umbilical trocar level with subsequent application of AGHO depending on the randomization performed.
  Arms: Group B. Solution hyperoxygenated fatty acids
Procedure: Physiological saline — The intervention consisted of placing a prosthesis at the umbilical trocar level with subsequent application of SSF depending on the randomization performed.
  Arms: Group A. Physiological saline.

SUMMARY:
TITLE:

Application of hyperoxygenated fatty acids (PrevOmega) in a surgical wound of the umbilical trocar after laparoscopic cholecystectomy with placement of prostheses in patients with risk factors.

OBJECTIVE: This study aimed to evaluate the effect of topical application of hyperoxygenated fatty acids (AGHO), PrevOmega, at the umbilical trocar level after laparoscopic cholecystectomy with prosthesis placement, regarding its non-application, on the infection rate. of the surgical site (ISQ) and eventration of the trocar orifice (EOT), in patients with risk factors for ISQ AND EOT.

METHODS: A prospective, double-blind, randomized study was performed in patients operated on for scheduled cholelithiasis, who also had any of the following risk factors that increase the appearance of SSI or OOT: BMI> 30kg / m2, Diabetes Mellitus, age> 65 years and Chronic Obstructive Pulmonary Disease. Group A was administered physiological saline (SSF) at the umbilical trocar level at the end of the intervention versus the administration of PrevOmega to group B. The study was carried out between January 2018 and January 2020 and is registered in the European Database of Clinical Trials with the EudraCT Code: 2018-002260-67.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of topical application of hyperoxygenated fatty acids (AGHO), PrevOmega, at the umbilical trocar level after laparoscopic cholecystectomy with prosthesis placement, regarding its non-application, on the infection rate. of the surgical site (ISQ) and eventration of the trocar orifice (EOT), in patients with risk factors for ISQ AND EOT.

ELIGIBILITY:
Inclusion Criteria:

Patients with ages between 18 and 90 years who underwent elective laparoscopic cholecystectomy for symptomatic cholelithiasis and who also presented any of the following risk factors for SSI or EOT were included:

* Obesity with body mass index (BMI)> 30kg / m2
* Diabetes Mellitus (insulin dependent or oral antidiabetic takers)
* Age (> 65 years)
* Chronic Obstructive Pulmonary Disease (COPD in treatment with inhalers).

Exclusion Criteria:

* Non-compliance with the inclusion criteria
* Conversion to laparotomy during the intervention
* Non-acceptance by the patient to participate in the study,
* Loss to follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2020-01-04 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 1 year
  Surgical site infection rate in patients with risk factors for infection and eventration after laparoscopic cholecystectomy

SECONDARY OUTCOMES:
Trocar hole eventration | 1 year
  Trocar hole eventration rate in patients with risk factors for infection and eventration after laparoscopic cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Laura Armañanzas, Study Director — HGUE
Locations (1):
- Marta, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowler PG, Jones SA, Walker M, Parsons D. Microbicidal properties of a silver-containing hydrofiber dressing against a variety of burn wound pathogens. J Burn Care Rehabil. 2004 Mar-Apr;25(2):192-6. doi: 10.1097/01.bcr.0000112331.72232.1b. PMID 15091147
- [Background] Chopra I. The increasing use of silver-based products as antimicrobial agents: a useful development or a cause for concern? J Antimicrob Chemother. 2007 Apr;59(4):587-90. doi: 10.1093/jac/dkm006. Epub 2007 Feb 16. PMID 17307768
- [Background] Sanders D, Lambie J, Bond P, Moate R, Steer JA. An in vitro study assessing the effect of mesh morphology and suture fixation on bacterial adherence. Hernia. 2013 Dec;17(6):779-89. doi: 10.1007/s10029-013-1124-5. Epub 2013 Jun 19. PMID 23780573
- [Background] Lai NM, Chaiyakunapruk N, Lai NA, O'Riordan E, Pau WS, Saint S. Catheter impregnation, coating or bonding for reducing central venous catheter-related infections in adults. Cochrane Database Syst Rev. 2016 Mar 16;3(3):CD007878. doi: 10.1002/14651858.CD007878.pub3. PMID 26982376
- [Background] Fernandez-Gutierrez M, Olivares E, Pascual G, Bellon JM, San Roman J. Low-density polypropylene meshes coated with resorbable and biocompatible hydrophilic polymers as controlled release agents of antibiotics. Acta Biomater. 2013 Apr;9(4):6006-18. doi: 10.1016/j.actbio.2012.12.012. Epub 2012 Dec 20. PMID 23261925
- [Background] Tang Y, Zhang MJ, Hellmann J, Kosuri M, Bhatnagar A, Spite M. Proresolution therapy for the treatment of delayed healing of diabetic wounds. Diabetes. 2013 Feb;62(2):618-27. doi: 10.2337/db12-0684. Epub 2012 Oct 5. PMID 23043160
- [Background] Armananzas L, Ruiz-Tovar J, Arroyo A, Garcia-Peche P, Armananzas E, Diez M, Galindo I, Calpena R. Prophylactic mesh vs suture in the closure of the umbilical trocar site after laparoscopic cholecystectomy in high-risk patients for incisional hernia. A randomized clinical trial. J Am Coll Surg. 2014 May;218(5):960-8. doi: 10.1016/j.jamcollsurg.2014.01.049. Epub 2014 Feb 18. PMID 24680572
- [Background] Comajuncosas J, Vallverdu H, Orbeal R, Pares D. [Trocar site incisional hernia in laparoscopic surgery]. Cir Esp. 2011 Feb;89(2):72-6. doi: 10.1016/j.ciresp.2010.08.007. Epub 2011 Jan 20. Spanish. PMID 21255770
- [Background] Muysoms FE, Antoniou SA, Bury K, Campanelli G, Conze J, Cuccurullo D, de Beaux AC, Deerenberg EB, East B, Fortelny RH, Gillion JF, Henriksen NA, Israelsson L, Jairam A, Janes A, Jeekel J, Lopez-Cano M, Miserez M, Morales-Conde S, Sanders DL, Simons MP, Smietanski M, Venclauskas L, Berrevoet F; European Hernia Society. European Hernia Society guidelines on the closure of abdominal wall incisions. Hernia. 2015 Feb;19(1):1-24. doi: 10.1007/s10029-014-1342-5. Epub 2015 Jan 25. PMID 25618025
- [Background] Mangram AJ. A brief overview of the 1999 CDC Guideline for the Prevention of Surgical Site Infection. Centers for Disease Control and Prevention. J Chemother. 2001 Nov;13 Spec No 1(1):35-9. doi: 10.1179/joc.2001.13.Supplement-2.35. PMID 11936376
- [Background] Anderson DJ, Podgorny K, Berrios-Torres SI, Bratzler DW, Dellinger EP, Greene L, Nyquist AC, Saiman L, Yokoe DS, Maragakis LL, Kaye KS. Strategies to prevent surgical site infections in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Sep;35 Suppl 2:S66-88. doi: 10.1017/s0899823x00193869. No abstract available. PMID 25376070
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists; Infectious Disease Society of America; Surgical Infection Society; Society for Healthcare Epidemiology of America. Clinical practice guidelines for antimicrobial prophylaxis in surgery. Am J Health Syst Pharm. 2013 Feb 1;70(3):195-283. doi: 10.2146/ajhp120568. No abstract available. PMID 23327981
- [Background] Magill SS, Edwards JR, Bamberg W, Beldavs ZG, Dumyati G, Kainer MA, Lynfield R, Maloney M, McAllister-Hollod L, Nadle J, Ray SM, Thompson DL, Wilson LE, Fridkin SK; Emerging Infections Program Healthcare-Associated Infections and Antimicrobial Use Prevalence Survey Team. Multistate point-prevalence survey of health care-associated infections. N Engl J Med. 2014 Mar 27;370(13):1198-208. doi: 10.1056/NEJMoa1306801. PMID 24670166
- [Background] Ban KA, Minei JP, Laronga C, Harbrecht BG, Jensen EH, Fry DE, Itani KM, Dellinger EP, Ko CY, Duane TM. American College of Surgeons and Surgical Infection Society: Surgical Site Infection Guidelines, 2016 Update. J Am Coll Surg. 2017 Jan;224(1):59-74. doi: 10.1016/j.jamcollsurg.2016.10.029. Epub 2016 Nov 30. No abstract available. PMID 27915053
- [Background] Leaper DJ, Edmiston CE. World Health Organization: global guidelines for the prevention of surgical site infection. J Hosp Infect. 2017 Feb;95(2):135-136. doi: 10.1016/j.jhin.2016.12.016. Epub 2016 Dec 24. No abstract available. PMID 28139389
- [Background] Brathwaite S, Latchana N, Esemuede I, Harzman A, Husain S. Risk Factors for Surgical Site Infection in Open and Laparoscopic Hartmann Closure: A Multivariate Analysis. Surg Laparosc Endosc Percutan Tech. 2017 Feb;27(1):51-53. doi: 10.1097/SLE.0000000000000365. PMID 28145967
- [Background] Rangel-Huerta OD, Aguilera CM, Mesa MD, Gil A. Omega-3 long-chain polyunsaturated fatty acids supplementation on inflammatory biomakers: a systematic review of randomised clinical trials. Br J Nutr. 2012 Jun;107 Suppl 2:S159-70. doi: 10.1017/S0007114512001559. PMID 22591890
- [Background] Hidalgo MP, Ferrero EH, Ortiz MA, Castillo JM, Hidalgo AG. Incisional hernia in patients at risk: can it be prevented? Hernia. 2011 Aug;15(4):371-5. doi: 10.1007/s10029-011-0794-0. Epub 2011 Feb 12. PMID 21318557
- [Background] El-Khadrawy OH, Moussa G, Mansour O, Hashish MS. Prophylactic prosthetic reinforcement of midline abdominal incisions in high-risk patients. Hernia. 2009 Jun;13(3):267-74. doi: 10.1007/s10029-009-0484-3. Epub 2009 Mar 5. PMID 19262985
- [Background] Moreno-Sanz C, Picazo-Yeste JS, Manzanera-Diaz M, Herrero-Bogajo ML, Cortina-Oliva J, Tadeo-Ruiz G. Prevention of trocar site hernias: description of the safe port plug technique and preliminary results. Surg Innov. 2008 Jun;15(2):100-4. doi: 10.1177/1553350608318789. PMID 18492730
- [Background] Tonouchi H, Ohmori Y, Kobayashi M, Kusunoki M. Trocar site hernia. Arch Surg. 2004 Nov;139(11):1248-56. doi: 10.1001/archsurg.139.11.1248. PMID 15545574
- [Background] Desbois AP, Lawlor KC. Antibacterial activity of long-chain polyunsaturated fatty acids against Propionibacterium acnes and Staphylococcus aureus. Mar Drugs. 2013 Nov 13;11(11):4544-57. doi: 10.3390/md11114544. PMID 24232668
- [Background] Mil-Homens D, Bernardes N, Fialho AM. The antibacterial properties of docosahexaenoic omega-3 fatty acid against the cystic fibrosis multiresistant pathogen Burkholderia cenocepacia. FEMS Microbiol Lett. 2012 Mar;328(1):61-9. doi: 10.1111/j.1574-6968.2011.02476.x. Epub 2012 Jan 6. PMID 22150831
- [Background] McCullough MC, Chu CK, Duggal CS, Losken A, Carlson GW. Antibiotic Prophylaxis and Resistance in Surgical Site Infection After Immediate Tissue Expander Reconstruction of the Breast. Ann Plast Surg. 2016 Nov;77(5):501-505. doi: 10.1097/SAP.0000000000000275. PMID 25003455
- [Background] Cattoir V. Mechanisms of Antibiotic Resistance. 2016 Feb 10. In: Ferretti JJ, Stevens DL, Fischetti VA, editors. Streptococcus pyogenes: Basic Biology to Clinical Manifestations [Internet]. Oklahoma City (OK): University of Oklahoma Health Sciences Center; 2016-. Available from http://www.ncbi.nlm.nih.gov/books/NBK333414/ PMID 26866217
- [Background] Frieri M, Kumar K, Boutin A. Antibiotic resistance. J Infect Public Health. 2017 Jul-Aug;10(4):369-378. doi: 10.1016/j.jiph.2016.08.007. Epub 2016 Sep 6. PMID 27616769
- [Background] Minar E, Schillinger M. Innovative technologies for SFA occlusions: drug coated balloons in SFA lesions. J Cardiovasc Surg (Torino). 2012 Aug;53(4):481-6. PMID 22854528
- [Background] Meaume S, Colin D, Barrois B, Bohbot S, Allaert FA. Preventing the occurrence of pressure ulceration in hospitalised elderly patients. J Wound Care. 2005 Feb;14(2):78-82. doi: 10.12968/jowc.2005.14.2.26741. PMID 15739656
- [Result] Maicas VT, Rochina IJ. [Linoleic acid emulsion on the peri-lesion skin of venal ulcers. Action and cicatrizant effect. Corpus study]. Rev Enferm. 2008 Apr;31(4):26-32. Spanish. PMID 18564784